CLINICAL TRIAL: NCT01833884
Title: Hodgkin's Lymphoma: Prognostic Value of the Kinetic of Decrease of 5 Cytokines Concentration During Treatment
Brief Title: Kinetic of Cytokines Decrease and Hodgkin Lymphoma Prognostic
Acronym: CYTOKINES-LH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHB 09-02; RCB : 2009-A01117-50 (Other: AFSSAPS)
Record Dates: First submitted 2012-10-23; First posted 2013-04-17 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hodgkin's Disease
Keywords: Hodgkin Lymphoma, Adult; Cytokines; TARC; IL-6; IL1-RA; sCD30; TNFR1
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): Collection of blood specimen for Cytokines dosing scheduled before, during and after treatment of Hodgkin's lymphoma (last collection date about 90 days after the end of treatment)
  Interventions: Other: Collection of blood specimen

INTERVENTIONS:
Other: Collection of blood specimen — Collection of blood specimen for Cytokines dosing scheduled before , during and after treatment of Hodgkin's lymphoma (last collection date about 90 days after the end of treatment)

SUMMARY:
More than 90% of patients with Hodgkin lymphoma (HL) can recover thanks to conventional polychemotherapy regimens - ABVD or BEACOPP - with or without radiotherapy. Nevertheless, some patients relapse and others are resistant to any treatment. These patients represent 2-5% of stage I / II and 5-10% of disseminated stages. The usual prognostic index based on clinical and biological data (supradiaphragmatic HL: EORTC and advanced HL International Prognostic Score) cannot always detect patients at risk.

New prognostic factors are required to screen out these high risk patients. Among available biological factors, we will retain the cytokines secreted by tumor cells and cells from the environment.

Indeed, the prognostic value of plasma cytokines levels and their soluble receptors has recently been described by at least two teams. Olivier CASASNOVAS set up a prognostic index based on quantities of IL-1 RA, IL-6, sCD30 and TNFR1 at diagnosis,and the V. Diehl team published the prognostic value of the decrease of TARC (CC Thymus and Activation-related chemokine).

In daily practice, the early assessment of response by PET CT-scan is now an undeniable prognostic factor. Early identification of no-response or relapse is, in fact, based on clinical and imaging (PET-CT scan).

We propose to evaluate the decrease of cytokines concentration with a prognostic value (TARC, IL-6, IL1-RA, sCD30, TNFR1) as markers of response during treatment and during early follow-up. The dosage of these cytokines will be paired with radiological assessments.

A correlation between the decrease of cytokines plasma levels overtime and event-free survival will be searched afterwards.

DETAILED DESCRIPTION:
To evaluate the decrease of cytokines concentration with a prognostic value as markers of response, the dosage of TARC, IL-6, IL1-RA, sCD30 and TNFR1 will be performed during treatment at :diagnosis, cycle 1 day 15, cycle 2 Day 1, cycle 3 Day 1, Day 1 of consolidation (Cycle 5 day 1 or before radiotherapy) and evaluation of end of treatment.

an early follow-up with a dosage of cytokines will be performed 3 months after the end of treatment.

An evaluation for Event Free Survival will be done at 3 years from diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin Lymphoma diagnosis
* I-II or III-IV Stages
* untreated Patient (including corticosteroids)
* Patient treated and followed exclusively in center Henri Becquerel
* Informed Consent signed

Exclusion Criteria:

* psychological, social or family conditions not allowing a suitable follow-up for study
* Mental deficiency not allowing the good understanding of study procedures
* positive HIV serology
* positive B or C Hepatitis serology
* Pregnant or lactating
* Patient registered with a social security scheme or in an equivalent situation
* Patient in a period of exclusion on another biomedical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Decrease of cytokines concentration TARC, IL-6, IL1-RA, sCD30, TNFR1) as markers of response during treatment and during early follow-up in Hodgkin's disease | 90 days after end of treatment
  evaluate the decrease of cytokines concentration with a prognostic value (TARC, IL-6, IL1-RA, sCD30, TNFR1) as markers of response during treatment (At Cycle 1 Day 15 of chemotherapy,Cycle 2 Day 1, cycle 3 Day 1, Cycle 5 Day 1 or Day 1 of Radiotherapy, 1 month after the end of treatment) , and during early follow-up (3 months after the end of treatment) in patients with Hodgkin's disease

SECONDARY OUTCOMES:
Correlation between the decrease of cytokines plasma levels and event-free survival | 3 years
  Evaluation of correlation between the decrease of cytokines plasma levels and event-free survival after 3 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Aspasia STAMATOULLAS, MD, Principal Investigator — CENTRE HENRI BECQUEREL-Rouen
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No